CLINICAL TRIAL: NCT00237926
Title: Comparing Aerobic to Resistance Training in Recovery From Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriService Nursing Research Program (Other)
Responsible Party: Stacey Young-McCaughan, The Geneva Foundation at Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: N05-006
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Neoplasms
Keywords: Sleep; Fatigue; Exercise tolerance; Quality of life; Health status
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): aerobic exercise
  Interventions: Behavioral: Exercise
- 2 (Experimental): Resistance Training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — aerobic or resistance training

SUMMARY:
The purpose of this study is to compare the health outcomes of a 12-week exercise program focused on aerobic training (using a treadmill) to a 12-week exercise program focused on resistance training (using Thera-Bands) in sedentary patients within 6 months of completing treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* have a biopsy-proven cancer diagnosis
* be within six months of having completed chemotherapy or radiation therapy for treatment for cancer as determined by the primary physician
* be ambulatory but sedentary (i. e., has not followed an exercise regimen of a minimum of 3 times per week for at least 20 minutes each session over the previous six weeks)
* have an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 asymptomatic) or 1 (symptomatic, fully ambulatory)
* be at least 18 years old
* be able to read and speak English
* have a medical statement from either the patient's primary care provider or the primary oncologist indicating that participation in the program is not medically contraindicated

Exclusion Criteria:

* following an exercise regimen a minimum of 3 times per week for at least 20 minutes each session within the previous 6 weeks
* bone or joint destruction that could be aggravated with exercise
* severe cognitive impairment identified by either the patient's medical care provider or by the study team
* neuropathy-sensory common toxicity criteria (CTC) grade 3 (sensory loss or paresthesia interfering with activities of daily living) or grade 4 (permanent sensory loss that interferes with function) peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
quality of life | 12-weeks

SECONDARY OUTCOMES:
exercise tolerance | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Young-McCaughan, RN, PhD, Principal Investigator — United States Department of Defense
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States